CLINICAL TRIAL: NCT01005446
Title: PS-901: Prospective Multicenter Open Label Study of the Encore Reverse® Shoulder Prosthesis
Brief Title: Reverse Shoulder Prosthesis Prospective Multi-Center Study
Status: Completed | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: PS - 901
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Rotator Cuff Deficiency; Shoulder Arthropathy; Failed Shoulder Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RSP Device: Post Market Study
  Interventions: Device: Encore Reverse Shoulder Prosthesis (RSP®)

INTERVENTIONS:
Device: Encore Reverse Shoulder Prosthesis (RSP®) — The RSP is indicated for use in subjects with grossly rotator cuff deficient shoulder joints with severe arthropathy or a previously failed joint replacement with a grossly rotator cuff deficient shoulder joint.
  Other Names: RSP®

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the Reverse® Shoulder Prosthesis for treatment of rotator cuff deficiency in subjects who are candidates for a total shoulder replacement (primary and revision subjects).

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty for the treatment of rotator cuff deficiency and glenohumeral arthritis have shown favorable outcomes in pain and function over the short and medium term. A prospective, multi-center study on the outcomes of subjects treated with the RSP would be a valuable addition to the literature and give important information regarding an ever-increasing treatment option for subjects with rotator cuff deficiency. The study will take place at multiple sites across the United States and will be managed by the DJO Surgical Clinical Affairs Department. The study will include only subjects who meet the indications for use criteria for the Reverse® Shoulder Prosthesis and who are candidates for total shoulder replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a total shoulder joint replacement
* Subject must be diagnosed with one or more of the following conditions:

Irreparable rotator cuff tear with gleno-humeral arthritis; Failed rotator cuff surgery with gleno-humeral instability or antero- superior escape; Failed shoulder replacement surgery

* Subject has a functional deltoid muscle
* Subject's joint must be anatomically and functionally suited to receive the selected implant
* Subject is 60 years of age or older (≥ 60 yrs of age) at time of consent
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures
* Subject is not pregnant

Exclusion Criteria:

* Subject has a non-functional deltoid muscle
* Subject has a mental condition(s) that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is a prisoner
* Subject has high levels of physical activity (ex. competitive sports, heavy physical labor)
* Subject is pregnant
* Subject has an active infection or sepsis
* Subject has loss of ligamentous structures
* Subject has a history of alcoholism or other addictions (current or past)
* Subject has muscular, neurological or vascular deficiencies which compromise the affected extremity (i.e., Parkinson's Disease, Syringomyelia and Multiple Sclerosis, Charcot joints)
* Subject has severe glenoid bone loss
* Subject has known materials sensitivity (to metals)
* Subject is younger than 60 years of age (< 60 years of age) at consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are 60 years of age or older at the time of consent and are suffering from a grossly rotator cuff deficient shoulder joints with severe arthropathy or have a previously failed joint replacement with a grossly rotator cuff deficient shoulder joint.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2009-12; Primary Completion 2017-08 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Improvement in American Shoulder and Elbow Surgeons Score (ASES) from Baseline | 2 year
  Improvement in American Shoulder and Elbow Surgeons Score (ASES) from Baseline. Assessments include: 1) Pain score where 0=no pain at all and 10=pain as bad as it can be 2) Function score where 0=my should is useless and 10=my shoulder is normal 3) Activity score where 0=unable to do and 3=Normal.

SECONDARY OUTCOMES:
Radiologic Success | 5 year
  Changes in radiolucency compared with Baseline
Change in ASES score from Baseline | 5 year
  Improvement in American Shoulder and Elbow Surgeons Score (ASES) from Baseline. Assessments include: 1) Pain score where 0=no pain at all and 10=pain as bad as it can be 2) Function score where 0=my should is useless and 10=my shoulder is normal 3) Activity score where 0=unable to do and 3=Normal.
SF36- (Short Form 36)Health Survey | 5 year
  Change from baseline using the SF36-Health Status. There are multiple scales for general health, pain and activities of daily living
Change in Simple Shoulder Test from Baseline | 5 year
  Change in Simple Shoulder Test from Baseline. Twelve questions about pain and functionality with responses being yes or no
Subject Satisfaction Survey | 5 year
  Patient Related Outcome of Device Satisfaction (score 1-5 with 1 = best and 5 = worst) Device satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Samer S. Hasan, M.D., Principal Investigator — Cincinnati Sports Medicine and Orthopaedic Center
Locations (10):
- United States (10):
  - Stanford University - Dept. of Orthopedics, Redwood City, California
  - Coastal Orthopedics & Sports Medicine, Bradenton, Florida
  - Orthopaedic Institute at Holy Cross Hospital, Fort Lauderdale, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Norton Orthopaedic & Sports Medicine Specialists, Louisville, Kentucky
  - Excelsior Orthopaedics, Amherst, New York
  - Cincinnati Sports Medicine and Orthopeadic Center, Cincinnati, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Texas Center for Joint Replacement, Plano, Texas
  - Rimrock Orthopedics, St. George, Utah

REFERENCES:
- See also: Sponsor website — http://www.djosurgical.com